CLINICAL TRIAL: NCT02042027
Title: Subconjunctival IVIg (Gamunex-C) Injection for Corneal Neovascularization and Inflammatory Conditions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Balamurali Ambati, Professor of Ophthalmology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMB70983
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Corneal Neovascularization; Corneal Graft Failure; Anterior Segment Inflammation
Keywords: corneal neovascularization; Gamunex-C; IVI-g; anterior segment inflammation
MeSH Terms: conditions — Corneal Neovascularization | interventions — Hizentra; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Gamunex-C 50 mg subconjunctival injections, in addition to standard of care treatment (steroids and cyclosporine). One dose of Gamunex-C injection delivered four weeks prior to corneal transplant surgery and one dose at the time of corneal transplantation. Dose to be repeated if recurrence of corneal neovascularization
  Interventions: Drug: Gamunex-C
- Group B (Active Comparator): Gamunex-C 50 mg subconjunctival injections, one dose injected for patients with active disease from corneal melts (peripheral ulcerative keratitis; Mooren's ulcer), ocular cicatricial pemphigoid, or anterior uveitis refractory to conventional therapy.
  Interventions: Drug: Gamunex-C

INTERVENTIONS:
Drug: Gamunex-C — Patients will receive 50 mg (0.5 mL) subconjunctival Gamunex-C injection in addition to standard of care treatment (steroids and cyclosporine)
  Other Names: IVIg

SUMMARY:
The purpose of the study is to test the investigational drug Gamunex-C on the growth of blood vessels over the cornea. This study is being conducted by Dr. Balamurali Ambati at the Moran Eye Center at the University of Utah.

The cornea is the clear outer front part of the eye. In corneal neovascularization, blood vessels grow over the cornea. Corneal neovascularization and ocular anterior segment inflammations are sight-threatening conditions. Lipid deposition and edema with subsequent scar formation can compromise corneal clarity irreversibly. Corneal neovascularization is also a well recognized risk factor for corneal graft failure. In its natural state, the cornea is a site of immune privilege well suited to tissue transplantation. Once vascularized, there is direct exposure of corneal antigens to circulating host immune mechanisms greatly increasing the chance of rejection [Collaborative Corneal Transplantation Study].

Melting or inflammation in the anterior chamber, cornea, or ocular surface can cause irreversible scarring or destruction of the optical elements of the eye, which can compromise vision.

Current standard of care for such conditions includes use of topical steroids and sometimes immunosuppressants (e.g., cyclosporine). These do not address a common underlying corneal neovascularization or melting.

This is a Phase 1 clinical trial of subconjunctival IVIg (Gamunex-C) injection for treatment of corneal neovascularization in the setting of corneal transplantation with neovascularization. Candidates for corneal transplantation with corneal neovascularization in one or more quadrants crossing more than 0.5mm over the limbus will be identified for inclusion in our study.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates for corneal transplantation (only one eye per patient would be enrolled)
2. Patients with corneal neovascularization in one or more quadrants crossing more than 1.0 mm over the limbus at time of enrollment in the study
3. Patients with refractory anterior uveitis, non-responding corneal melts, or non-responding ocular cicatricial pemphigoid
4. Willing and able to comply with clinic visits and study-related procedures
5. Provide signed informed consent
6. Age 18 or over

Exclusion Criteria:

1. Patients receiving antiangiogenic anti-VEGF medication either systemically or intravitreally for other pathology or who have received these drugs within 3 months of study enrollment
2. Patients with active corneal infection requiring additional treatment modalities
3. Patients receiving coumadin with INR >2.0, other anti-thrombotic agents (e.g., aspirin, Plavix) permitted at discretion of investigator
4. History of CVA or MI within 6 months prior to study enrollment
5. Uncontrolled BP- defined as SBP>160 mmHg or DBP >95mmHg while patient is sitting
6. Pregnant or breast-feeding women
7. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Ability to regress neovascularization | at time of transplant
  Ability of subconjunctival IVIg (Gamunex-C) injection to regress neovascularization and promote graft survival after corneal transplantation, or retard corneal/anterior segment inflammation in patients with progressive/refractory conditions (corneal melts, ocular cicatricial pemphigoid, or refractory anterior uveitis)

SECONDARY OUTCOMES:
Ability to regress neovascularization and promote graft survival | 28 weeks after transplant
  ability of subconjunctival IVIg (Gamunex-C) injection to regress neovascularization and promote graft survival after corneal transplantation, or retard corneal/anterior segment inflammation in patients with progressive/refractory conditions (corneal melts, ocular cicatricial pemphigoid, or refractory anterior uveitis)
Ability to regress neovascularization and promote graft survival | 52 weeks after transplant
  ability of subconjunctival IVIg (Gamunex-C) injection to regress neovascularization and promote graft survival after corneal transplantation, or retard corneal/anterior segment inflammation in patients with progressive/refractory conditions (corneal melts, ocular cicatricial pemphigoid, or refractory anterior uveitis)
Need for immunosuppression | week 28
  need for immunosuppression at weeks 28 in both treatment groups
Need for immunosuppression | week 52
  need for immunosuppression at week 52 in both treatment groups
Effect on corneal infections | week 28
  Effect on corneal infections or other side effects through week 28 in both treatment groups
Effect on corneal infections | Week 52
  effect on corneal infections or other side effects through week 52 in both treatment groups
Visual outcome at week 28 | Week 28
  visual outcome (by ETDRS chart) at week 28 in both treatment groups
Visual outcome at week 52 | Week 52
  visual outcome (by ETDRS chart) at week 52 in both treatment groups
Mean number of injections through week 28 | week 28
  mean number of injections performed per patient through weeks 28
Mean number of injections through week 52 | week 52
  mean number of injections performed per patient through week 52 in patients receiving subconjunctival IVIg (Gamunex-C) injections
Need for rescue treatment in standard of care group | Week 28
  need for rescue treatment in the standard of care group through week 28
Need for rescue treatment in standard of care group | week 52
  need for rescue treatment in the standard of care group through week 52

CONTACTS AND LOCATIONS:
Overall Officials: Balamurali K Ambati, M.D., Ph.D., M.B.A., Principal Investigator — University of Utah
Locations (1):
- John A. Moran Eye Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Chang JH, Garg NK, Lunde E, Han KY, Jain S, Azar DT. Corneal neovascularization: an anti-VEGF therapy review. Surv Ophthalmol. 2012 Sep;57(5):415-29. doi: 10.1016/j.survophthal.2012.01.007. PMID 22898649
- [Background] Chang JH, Gabison EE, Kato T, Azar DT. Corneal neovascularization. Curr Opin Ophthalmol. 2001 Aug;12(4):242-9. doi: 10.1097/00055735-200108000-00002. PMID 11507336
- [Background] Cho YK, Uehara H, Young JR, Tyagi P, Kompella UB, Zhang X, Luo L, Singh N, Archer B, Ambati BK. Flt23k nanoparticles offer additive benefit in graft survival and anti-angiogenic effects when combined with triamcinolone. Invest Ophthalmol Vis Sci. 2012 Apr 30;53(4):2328-36. doi: 10.1167/iovs.11-8393. PMID 22427553
- [Background] Singh SR, Grossniklaus HE, Kang SJ, Edelhauser HF, Ambati BK, Kompella UB. Intravenous transferrin, RGD peptide and dual-targeted nanoparticles enhance anti-VEGF intraceptor gene delivery to laser-induced CNV. Gene Ther. 2009 May;16(5):645-59. doi: 10.1038/gt.2008.185. Epub 2009 Feb 5. PMID 19194480
- [Background] Jani PD, Singh N, Jenkins C, Raghava S, Mo Y, Amin S, Kompella UB, Ambati BK. Nanoparticles sustain expression of Flt intraceptors in the cornea and inhibit injury-induced corneal angiogenesis. Invest Ophthalmol Vis Sci. 2007 May;48(5):2030-6. doi: 10.1167/iovs.06-0853. PMID 17460257
- [Background] Luo L, Zhang X, Hirano Y, Tyagi P, Barabas P, Uehara H, Miya TR, Singh N, Archer B, Qazi Y, Jackman K, Das SK, Olsen T, Chennamaneni SR, Stagg BC, Ahmed F, Emerson L, Zygmunt K, Whitaker R, Mamalis C, Huang W, Gao G, Srinivas SP, Krizaj D, Baffi J, Ambati J, Kompella UB, Ambati BK. Targeted intraceptor nanoparticle therapy reduces angiogenesis and fibrosis in primate and murine macular degeneration. ACS Nano. 2013 Apr 23;7(4):3264-75. doi: 10.1021/nn305958y. Epub 2013 Mar 20. PMID 23464925